CLINICAL TRIAL: NCT02078908
Title: The Effect of Sodium Nitrite on Renal Variables, Brachial and Central Blood Pressure in Healthy Humans. A Randomized, Cross Over, Placebo Controlled Dose-response Study
Brief Title: The Effect of Sodium Nitrite on Renal Function and Blood Pressure in Healthy Humans. A Dose-response Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Chief physician, PhD, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: JBR-1-2013; 2013-002211-10 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2014-03-05 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Central blood pressure; Peripheral (brachial) blood pressure; Renal variables; Vasoactive hormones; Pharmacology; Pharmacokinetics
MeSH Terms: interventions — Sodium Nitrite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 40 micrograms sodium nitrite (Active Comparator): Continuous 2 hour infusion of sodium nitrite, 40 micrograms/kg/hour
  Interventions: Drug: Sodium nitrite, 40 micrograms/kg/hour
- 120 micrograms sodium nitrite (Active Comparator): Continuous 2 hour infusion of sodium nitrite, 120 micrograms/kg/hour
  Interventions: Drug: Sodium nitrite, 120 micrograms/kg/hour
- 240 micrograms sodium nitrite (Active Comparator): Continuous 2 hour infusion of sodium nitrite, 240 micrograms/kg/hour
  Interventions: Drug: Sodium nitrite, 240 micrograms/kg/hour
- Placebo (Placebo Comparator): Continuous 2 hour infusion of sodium chloride, 25 ml/hour
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium nitrite, 40 micrograms/kg/hour — Continuous 2 hour infusion of sodium nitrite, 40 micrograms/kg/hour
  Other Names: NaNO2; ATC V03AB08; EV substance code: SUB15308MIG; CAS15 number: 7632-00-0
  Arms: 40 micrograms sodium nitrite
Drug: Sodium nitrite, 120 micrograms/kg/hour — Continuous 2 hour infusion of sodium nitrite, 120 micrograms/kg/hour
  Other Names: NaNO2; ATC V03AB08; EV substance code: SUB15308MIG; CAS15 number: 7632-00-0
  Arms: 120 micrograms sodium nitrite
Drug: Sodium nitrite, 240 micrograms/kg/hour — Continuous 2 hour infusion of sodium nitrite, 240 micrograms/kg/hour
  Other Names: NaNO2; ATC V03AB08; EV substance code: SUB15308MIG; CAS15 number: 7632-00-0
  Arms: 240 micrograms sodium nitrite
Drug: Placebo — Continuous 2 hour infusion of sodium chloride, 25 ml/hour
  Other Names: Sodium chloride
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of different doses of sodium nitrite infusion in 12 healthy subjects. The effects on renal handling of nitrite, nitrate, sodium and water, plasma concentrations of vasoactive hormones, peripheral (brachial) and central blood pressure will be evaluated.

Hypothesis

Sodium nitrite infusion

1. increases urinary sodium excretion and renal filtration rate
2. lowers blood pressure, central as well as peripheral
3. affects vasoactive hormones
4. it is possible to establish a dose that affects the renal function with only minor effect on the blood pressure.

DETAILED DESCRIPTION:
Background:

Nitric oxide (NO) is an important vasodilating molecule with a very complex biochemistry and metabolism. NO is classically synthesized from L-arginin by endothelial nitric oxide synthase (eNOS) located in the endothelial cell lining. Several chronic cardiovascular diseases such as hypertension, chronic kidney disease and diabetes are accompanied by endothelial dysfunction and hence diminished synthesis of NO. NO is a very reactive molecule and direct investigation of its function are limited and it has mainly been investigated by inhibition of eNOS. Recent research has shown that sodium nitrite is readily converted to NO by enzymes in vivo. The effects of sodium nitrite on renal variables, vasoactive hormones and central blood pressure are previously unexamined. It is now possible to achieve serial estimations of the central aortic systolic pressure (CASP) by newly designed wrist born device.

Hypothesis:

1. Sodium nitrite infusion increases the urinary sodium excretion and glomerular filtration rate (GFR) in a dose related manner.
2. Sodium nitrite infusion increases plasma levels of nitrite, nitrate, NO and cyclic guanosine monophosphate (cGMP)
3. Sodium nitrite infusion lowers the peripheral and central blood pressure
4. Renal clearance of nitrite is constant and not dose dependent
5. Sodium nitrite infusion affects vasoactive hormones
6. It is possible to establish a dose that affects the renal variables with only minor effect on the blood pressure.

Purpose:

The purpose of this study is to investigate the effects of sodium nitrite infusion on

1. Renal handling of nitrite, nitrate, sodium and water
2. Plasma concentrations of vasoactive hormones
3. Peripheral (brachial) blood pressure and CASP

Design:

12 healthy subjects are recruited in this randomised, cross over, placebo controlled, single-blinded study. Each subject will attend to four examination days. Four days prior to each examination day subjects are given a standardized diet with a low level of nitrate and nitrite. On the evening before the examination day the subjects take a single dose of lithium carbonate 300 mg in order to measure lithium clearance. On the examination days subjects are receiving a two hour infusion of either placebo (isotonic sodium chloride) or one of three doses of sodium nitrite. During the four examination days each subject receives all treatments in random order.

Perspectives:

Knowledge regarding hemodynamic and renal dose-response relationship is essential, in order to carry out future planned studies of the nitrite-NO system, in hypertensive subjects and during simultaneous modulation of various enzyme systems, involved in the conversion of nitrite to NO. Increasing knowledge about the nitrite-NO system can contribute to changing the clinical practise of diagnostics and treatment of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18,5-30 kg/m2
* Women must use safe contraception

Exclusion Criteria:

* Tobacco smoking, medicine or substance abuse
* Weekly consumption of more than 21 standard drinks of alcohol for men and 14 standard drinks of alcohol for women (1 danish standard drink equals 12 grams of alcohol)
* Medical treatment in the last 2 weeks except for contraception
* Pregnancy or nursing
* Diabetes mellitus
* estimated glomerular filtration rate (eGFR) < 60 ml/min
* neoplasm
* clinically significant heart, lung, liver, kidney, metabolic og neurologic disease
* clinically significant findings in screening blood samples, urine sample or ECG
* Office blood pressure > 140/90 mmHg
* Blood donation within 1 month of the first day of investigation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Fractional urinary sodium excretion | One day

SECONDARY OUTCOMES:
Nitrite clearance | One day
Nitrate clearance | One day
Glomerular filtration rate | One day
  Measured by determent renal clearance of 51Cr-EDTA (51-chrome ethylenediaminetetraacetic acid) using constant infusing technique
Proximal sodium transport | One day
  Proximal sodium transport is estimated by lithium clearance
Free water clearance | One day
Urinary excretion of cyclic guanosine monophosphate (cGMP) | One day
Urinary excretion of epithelial sodium channels (ENaC) | One day
Urinary excretion of water channels (aquaporin-2) | One day
Plasma concentration of renin | One day
Plasma concentration of angiotensin 2 | One day
Plasma concentration of aldosterone | One day
Plasma concentration of atrial natriuretic peptide (ANP) | One day
Plasma concentration of brain natriuretic peptide (BNP) | One day
Plasma concentration of cyclic guanosine monophosphate (cGMP) | One day
Plasma concentration of endothelin | One day
Plasma concentration of vasopressin (AVP, ADH) | One day
Peripheral (brachial) blood pressure | One day
  Measured by oscillometric sphygmomanometer, Omron 705IT, Omron Matsusaka CO. Ltd.
Central aortic systolic blood pressure (CASP) | One day
  Estimated by tonometric pulse wave analysis. Device: BPro from HealthSTATS International, Singapore

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, MD, PhD, Principal Investigator — Regional Hospital Holstebro
Locations (1):
- Department of Medical Research, Regional Hospital Holstebro, Holstebro, Denmark